CLINICAL TRIAL: NCT06849570
Title: Assessment of the PEEP Responsiveness to Titrate End-expiratory Pressure and of the Need for Muscle Relaxation During Prone Positioning in Moderate-to-severe Acute Respiratory Distress Syndrome: A Master Protocol
Acronym: PEPER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APHP240459
Record Dates: First submitted 2024-12-16; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Intensive Care Units (ICUs)
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Master Protocol, including two randomized, controlled, clinical trials with Bayesian adaptive designs
  * First randomization with 3 parallel arms (first ratio 1:1:1) A. Minimal distension B. Maximal recruitment C. PRT-guided ventilation strategy
  * Second randomization within 4 to 72 hours, if persistent PaO2/FiO2 ≤150 mmHg, with two parallel arms (ratio 1:1)
    1. Prone position with systematic NMBAs
    2. Prone position without systematic NMBAs
Who Masked: Care Provider, Investigator
Masking Description: Medical team blinded for first randomization. The second randomization is open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First randomization : Arm A : Routine care Minimal distention (Active Comparator): Decision of the ventilation strategy according to the routine care
  Interventions: Other: Minimal distension
- First randomization : Arm B Routine care maximal recruitment (Active Comparator): Decision of the ventilation strategy according to the routine care
  Interventions: Other: Maximal Recruitment
- First randomization: Arm C : Decision of th ventilation strategy according to the PRT result (Experimental): Maximal recruitment strategy in patients with positive PEEP responsiveness test (PRT) or minimal distension strategy in patients with negative PRT.
  Interventions: Other: Minimal distension; Other: Maximal Recruitment
- Second randomization : NMBAs used as a rescue (Active Comparator)
  Interventions: Other: Prone position + rescue NMBAs
- Second randomization : early NMBAs used as soon as possible (Experimental)
  Interventions: Other: Prone position + early NMBAs

INTERVENTIONS:
Other: Minimal distension — Patients receive tidal volume (VT) of 6 mL/kg and conservative positive end-expiratory pressure (PEEP) setting.
  Arms: First randomization : Arm A : Routine care Minimal distention; First randomization: Arm C : Decision of th ventilation strategy according to the PRT result
Other: Maximal Recruitment — Patients receive tidal volume adjusted to limit plateau pressure (∆P) to 14 cmH2O and the highest possible PEEP while maintaining plateau pressure (PPLAT) ≤ 27 cmH2O.
  Arms: First randomization : Arm B Routine care maximal recruitment; First randomization: Arm C : Decision of th ventilation strategy according to the PRT result
Other: Prone position + early NMBAs — NMBAs given as soon as possible after randomization
  Arms: Second randomization : early NMBAs used as soon as possible
Other: Prone position + rescue NMBAs — NMBAs given only as a rescue
  Arms: Second randomization : NMBAs used as a rescue

SUMMARY:
Despite best supportive care, mortality of the Acute Respiratory Distress Syndrom (ARDS) remains high. In the absence of specific treatments, providing safe and efficient mechanical ventilation (MV) is key to survival.

The use of low tidal volumes (VT) and plateau pressures (PPLAT) improves survival in randomized controlled trials (RCTs), but the safest VT to be applied for each patient remains unknown. Whether targeting low ∆P instead of a 6 mL/kg VT improves outcome has not been tested prospectively. The optimal method to set PEEP is also a matter of debate. As the amount of potentially recruitable lung vary widely among patients and is strongly associated with the response to PEEP, it may be necessary to tailor PEEP settings based on the response to a PEEP trial.

The first aim is to test a personalized approach to set PEEP widely supported by the literature. The first hypothesis is that i) patients with greater amounts of recruitable lung may benefit from higher PEEP levels, provided that attention is paid to maintain ∆P below 14 cmH2O, ii) setting PEEP based on results of a PEEP-responsiveness test improves survival as compared to low- and high-PEEP strategies applied independently of the patient response.

Apart from VT reduction and PPLAT control below 30 cmH2O, only 2 interventions demonstrated a reduction of mortality in large RCTs: a 48-hour continuous infusion of neuromuscular blocking agents (NMBAs) at the acute phase of ARDS6 and the use of prone positioning (PP). Whereas there is little doubt on the utility of PP in patients with PaO2/FiO2 ratio < 150 mmHg, there is more controversy on the impact of NMBAs on survival. Despite a strong rationale and a very widespread use in clinical practice, no current guidelines answer the question of the best timing of muscle relaxation in moderate to severe ARDS patients treated with PP.

As a second aim, the hypothesis is that the early systematic and combined use of NMBAs improved survival of patients with moderate to severe ARDS requiring prone positioning after optimization of PEEP settings.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation within 96 hours of ICU admission and within 72 hours of tracheal intubation for first randomization and then within 72 hours of the first randomization for the second randomization
* Patients meeting the Berlin ARDS definition criteria with hypoxemia characterized as

  * for first randomization: PaO2/FiO2 ≤150 mmHg on a PEEP ≥5 cmH2O with FiO2≥0.6 while VT is 6 ml/kg Predicted Body Weight (PBW) and adequate sedation level to adjust mechanical ventilation settings
  * for second randomization: PaO2/FiO2 ≤150 mmHg on optimized ventilatory settings according to the first randomization, confirmed by two Arterial blood gas (ABG) analyses separated by an interval time of 4 hours and observed within 72 hours of the first randomization
* Informed consent signed:

  * by the patient
  * Or informed consent signed by a family members/trustworthy person if his condition does not allow him to express his consent by written as per L. 1111-6
  * Or in a situation urgently and in the absence of family members/trustworthy person, the patient can be enrolled. The consent to participate to the research will be requested as soon as the condition of the patient will allow him to consent.
* Health insurance coverage

Exclusion Criteria:

* Age < 18 years
* Known pregnancy or breastfeeding
* Participation in another interventional studies as long as these studies do not interfere with the primary endpoint and the secondary safety objectives of PEPER, or being in the exclusion period at the end of a previous study.
* Intracranial pressure > 30 mm Hg or cerebral perfusion pressure < 60 mmHg
* Severe chronic respiratory disease requiring long-term O2 therapy or home mechanical ventilation (except Continuous positive arway pressure (CPAP)/ Bilevel positive airway pressure (BIPAP) used for sleep apnea syndrome)
* Chronic interstitial lung disease
* Continuous neuromuscular blockade infusion at enrolment
* Previous hypersensitivity or anaphylactic reaction to any NMBA
* Neuromuscular disease that may potentiate neuromuscular blockade or impair spontaneous ventilation: amyotrophic lateral sclerosis, Guillain-Barré syndrome, myasthenia gravis, upper spinal injury at level C5 or above
* Patients on ECMO or any technique of extracorporeal CO2 removal
* Sickle cell disease
* Actual body weight >1 kg/cm of height
* Severe chronic liver disease defined as a Child-Pugh score of 12-15
* Pneumothorax at randomization
* Expected duration of mechanical ventilation <48 hours
* Simplified acute physiology score SAPS II score >75 at the time of enrolment or suffering from a disease with an estimated survival time of less than two months
* Decision to withhold life-sustaining treatment
* Patients deprived of freedom or under legal authority
* Unstable spine fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days after randomization

SECONDARY OUTCOMES:
Ratio of arterial oxygen partial pressure to inspired oxygen fraction | 24 hours after randomization
  PaO2/FiO2
Ratio of arterial oxygen partial pressure to inspired oxygen fraction | 48 hours after randomization
  PaO2/FiO2
Ratio of arterial oxygen partial pressure to inspired oxygen fraction | 72 hours after randomization
  PaO2/FiO2
Ratio of arterial oxygen partial pressure to inspired oxygen fraction | 7 days after randomization
  PaO2/FiO2
Ratio of arterial oxygen partial pressure to inspired oxygen fraction | 14 days after randomization
  PaO2/FiO2
Oxygen index | 24 hours after randomization
Oxygen index | 48 hours after randomization
Oxygen index | 72 hours after randomization
Oxygen index | 7 days after randomization
Oxygen index | 14 days after randomization
Tidal volume | 24 hours after randomization
  Amount of air that is inhaled or exhaled during a normal, relaxed breath
Tidal volume | 48 hours after randomization
  Amount of air that is inhaled or exhaled during a normal, relaxed breath
Tidal Volume | 72 hours after randomization
  Amount of air that is inhaled or exhaled during a normal, relaxed breath
Tidal Volume | 7 days after randomization
Tidal Volume | 14 days after randomization
Respiratory Rate | 24 hours after randomization
Sequential Organ Failure Assessment (SOFA) score | 24 hours after randomization
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Sequential Organ Failure Assessment (SOFA) score | 48 hours after randomization
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Sequential Organ Failure Assessment (SOFA) score | 72 hours after randomization
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Sequential Organ Failure Assessment (SOFA) score | 7 days after randomization
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Sequential Organ Failure Assessment (SOFA) score | 14 days after randomization
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
All-cause mortality | 90 days after inclusion
All-cause mortality | 1 year after inclusion
All-cause Intensive care unit mortality | 90 days after inclusion
All-cause Intensive care unit mortality | 1 year after inclusion
All-cause hospital mortality | 90 days after inclusion
All-cause hospital mortality | 1 year after inclusion
Duration of mechanical ventilation | Up to 1 year
Ventilator Free Days | 28 days after inclusion
Intensive Care Unit length of stay | Up to 1 year
Hospital length of stay | Up to 1 year
ICU free-days | 28 days after inclusion
Respiratory Rate | 48 hours after randomization
Respiratory Rate | 72 hours after randomization
Respiratory Rate | 7 days after randomization
Respiratory Rate | 14 days after randomization
Total Postitive end-expiratory pressure (PEEP) | 24 hours after randomization
Total Positive end-expiratory pressure (PEEP) | 48 hours after randomization
Total Positive end-expiratory pressure (PEEP) | 72 hours after randomization
Total Positive end-expiratory pressure (PEEP) | 7 days after randomization
Total Positive end-expiratory pressure (PEEP) | 14 days after randomization
Peak Pressure | 24 hours after randomization
Peak Pressure | 48 hours after randomization
Peak Pressure | 72 hours after randomization
Peak Pressure | 7 days after randomization
Peak Pressure | 14 days after randomization
Plateau Pressure | 24 hours after randomization
Plateau Pressure | 48 hours after randomization
Plateau Pressure | 7 days after randomization
Plateau Pressure | 14 days after randomization
compliance of the respiratory system | 24 hours after randomization
compliance of the respiratory system | 48 hours after randomization
compliance of the respiratory system | 72 hours after randomization
compliance of the respiratory system | 7 days after randomization
compliance of the respiratory system | 14 days after randomization
Hospital-free-days | 28 days after inclusion
Hospital-free-days | 90 days after inclusion
Occurence of barotrauma | 7 days after inclusion
  Defined as any pneumothorax, subcutaneous emphysema, pneumomediastinum, or pneumatocele of more than 2 cm detected on image examinations
Occurrence of acute cor pulmonale | 7 days after inclusion
  Defined by the combination of a right/left ventricular diameter ratio greater than 0.6 and a paradoxical septum
ICU acquired weakness | Up to 1 year
  Assessed by the medical research council (MRC) score at ICU discharge. The score ranges from 0 to 60. A score < 48 defines ICU acquired weakness
Number of days using other rescue procedures | Up to 1 year
  Other rescue procedure including inhaled nitric oxide, almitrine, epoprostenol sodium, extracorporeal membrane oxygenation (ECMO), extracorporeal CO2 removal (ECCO2R)
Use of NMBAs during the first 3 days following the first randomization or following inclusion in the rescue arm of the second randomization | Up to day 28
Muscle relaxants-free days | Up to day 7
  Between inclusion and day 7
Number of days alive and without continuous IV administration of sedatives/analgesics | At day 7
Number of days alive and without continuous IV administration of sedatives/analgesics | At day 28
Presence of delirium (CAM-ICU) | At day 14
Presence of delirium (CAM-ICU) | Up to 1 year
  At ICU discharge
Disability | At 1 year
  Assessed by the Activities of Daily Living score (Lawton IADL) The score is divided in 8 domains and ranges from 0 to 8. The higher the score, the more independent is the person.
Quality of life questionnaire | At 1 year
  Using EQ-5D-5L It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Post-Traumatic Stress Disorder (PTSD) | At 1 year
  Using the Impact Event Scale-Revised (IES-R) It contains 22 items scored on a 5-point Likert scale Total score ranges from 0 to 88. Higher scores indicate more severe symptoms.
Cognitive dysfunction | At 1 year
  Using T-MoCA score It evaluates 8 cognitive domains. The total score ranges from 0 to 30 points. A score of 26 or higher is considered as normal.
Return to work status | At 1 year
  Subsequent return to work. Return to work status: employment status
Place of residence | At 1 year
Paralysis recall assessment | At 1 year
  Using a modified Brice questionnaire Patient responses are categorized into levels of awareness and analyzed to determine if awareness occured and its nature. The result can be : no awareness, awareness with explicit recall, awareness with dreams, emotional distress, inconclusive responses
Severe acidosis | Within 8 hours after randomization
  pH<7.10

OTHER OUTCOMES:
Death with refractory hypoxemia | Up to day 7
  Defined as PaO2/FiO2< 80 mmHg outside a care incident
Death with refractory acidosis | Up to day 7
  Defined as Ph<7.10 despite Respiratory Rate (RR) ≥ 35 /min & VT 8 ml/kg
Death with barotrauma | Up to day 7
Need of commencement or 30% increase in vasopressors or hypotension (MAP<60 mmHg) | Within 8 hours after randomization
Refractory hypoxemia | Within 8 hours after randomization
  Defined as PaO2/FiO2< 50 mmHg for more than one hour

IPD SHARING:
Plan to Share IPD: Undecided